CLINICAL TRIAL: NCT02172885
Title: Mesenchymal Stem Cell Based Therapy for the Treatment of Osteogenesis Imperfecta
Acronym: TERCELOI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital de Cruces (Other)
Collaborators: Hospital Universitario Getafe (Other); Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Responsible Party: Principal Investigator, Clara I. Rodríguez, PI Stem Cell Laboratory, Hospital de Cruces
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT Number:2012-002553-38; Health Department of Spain (Other Grant/Funding Number: EC10-219)
Record Dates: First submitted 2014-06-12; First posted 2014-06-24 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Osteogenesis Imperfecta
Keywords: Mesenchymal stem cell based therapy; cell infusion
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal stem cells (Experimental): Five Mesenchymal Stem Cell infusions
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — Mesenchymal Stem Cell Infusions

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of five infusions of characterized HLA-identical MSC in non immunosuppressed children with Osteogenesis Imperfecta (OI).

DETAILED DESCRIPTION:
The principal aim of this trial is to assess the safety of non-mutated HLA-identical Mesenchymal stem cell (MSC) transplantation for OI pediatric patients irrespective of treatment with biphosphonates. Since MSC are inherently non-immunogenic and do not elicit proliferation of allogeneic lymphocytes (in co-culture experiments), a cell therapy based on HLA-identical or histocompatible (at least 5 shared out of 6 HLA antigens) allogenic MSC may be accomplished without subjecting the patients to immunosuppressor treatment. Adverse secondary effects due to immunosuppressor treatment will be avoided using this strategy thus patients may benefit from two cellular infusions. The patients will be followed for 2 years post their fifth and last MSC infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient age: older than 6 months and younger than 12 years old.
* Patients with molecular confirmation of mutation in either COL1A1 or COL1A2 genes associated with OI (type III).
* Patients with HLA identical (that shared at least 5/6 antigens) siblings willing to donate bone marrow-MSCs.
* All patients that fulfil the inclusion criteria regardless of whether or not they are undergoing biphosphonate treatment.
* Patients whose parents or the legal guardians are willing to sign the consent forms to participate in this clinical trial.

Exclusion Criteria:

* Patient age: older than 12 years old
* Patients lacking confirmation of mutation in either COL1A1 or COL1A2 genes associated with severe deforming OI (type III).
* Other pathological subtypes of OI.
* Patients lacking of HLA identical (that shared at least 5/6 antigens) siblings willing to donate bone marrow-MSCs.
* Immunodeficiencies and any other malignancies.
* Participation in other clinical trial.
* Any medical or psychiatric condition that in the researcher´s opinion could affect the patient´s ability to complete the trial or hamper the participation in the trial.
* Patients whose parents or the legal guardians do not sign the consent forms

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2014-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events as a Measure of Safety | up to 2 years post last MSCs infusion

SECONDARY OUTCOMES:
bone mineral density | up to 2 years post last MSCs infusion
fracture rate | up to 2 years post last MSCs infusion
growth velocity | up to 2 years post last MSCs infusion
change from baseline in degree of functionality | up to 2 years post last MSCs infusion
  9 question survey using a Bleck functional scale
change from baseline in well-being | up to 2 years post last MSCs infusion
  A 20 item questionnaire designed to evaluate the well-being will be used

CONTACTS AND LOCATIONS:
Overall Officials: Clara I. Rodríguez, Ph. D., Principal Investigator — BioCruces Health Research Institute/Cruces University Hospital
Locations (2):
- Spain (2):
  - Hospital Universitario Cruces, Barakaldo, Bizkaia
  - Hospital Universitario Getafe, Getafe, Madrid

REFERENCES:
- [Background] Infante A, Gener B, Vazquez M, Olivares N, Arrieta A, Grau G, Llano I, Madero L, Bueno AM, Sagastizabal B, Gerovska D, Arauzo-Bravo MJ, Astigarraga I, Rodriguez CI. Reiterative infusions of MSCs improve pediatric osteogenesis imperfecta eliciting a pro-osteogenic paracrine response: TERCELOI clinical trial. Clin Transl Med. 2021 Jan;11(1):e265. doi: 10.1002/ctm2.265. PMID 33463067
- [Result] Infante A, Cabodevilla L, Gener B, Rodriguez CI. Circulating TGF-beta Pathway in Osteogenesis Imperfecta Pediatric Patients Subjected to MSCs-Based Cell Therapy. Front Cell Dev Biol. 2022 Feb 9;10:830928. doi: 10.3389/fcell.2022.830928. eCollection 2022. PMID 35223854
- See also: Reiterative infusions of MSCs improve pediatric osteogenesis imperfecta eliciting a pro-osteogenic paracrine response: TERCELOI clinical trial — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC7805402/

DOCUMENTS (1):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT02172885/Prot_000.pdf